CLINICAL TRIAL: NCT05375136
Title: A Post Marketing Surveillance Study of Lenvatinib in Combination With Pembrolizumab in Korean Patients
Brief Title: A Study of Lenvatinib in Combination With Pembrolizumab in Korean Patients
Status: Completed | Type: Observational
Sponsor: Eisai Korea Inc. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Other Study IDs: E7080-M065-513
Record Dates: First submitted 2022-05-10; First posted 2022-05-16 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2023-07

CONDITIONS: Endometrial Neoplasms; Endometrium; Carcinoma; Renal Cell Carcinoma
Keywords: Lenvatinib; Pembrolizumab
MeSH Terms: conditions — Endometrial Neoplasms; Carcinoma; Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- All Participants: Participants who are prescribed with lenvatinib/pembrolizumab combination per approved prescribing information of lenvatinib and pembrolizumab in the post marketing setting will be enrolled and observed for up to 48 weeks or until clinical benefit or unacceptable toxicity occurs or discontinuation of therapy due to any reason, whichever occurs first.
  Interventions: Other: Non-interventional

INTERVENTIONS:
Other: Non-interventional — No intervention will be administered.

SUMMARY:
The purpose of this study is to collect and evaluate the following information in relation to the safety and the efficacy of Lenvatinib in lenvatinib/pembrolizumab combination therapy in the post marketing setting: (1) Serious adverse events and serious adverse drug reactions (2) Unexpected adverse events and adverse drug reactions not reflected in the approved product package insert of lenvatinib in lenvatinib/pembrolizumab combination therapy (3) Known adverse drug reactions (4) Non-serious adverse drug reactions (5) Other safety and efficacy related information.

ELIGIBILITY:
Inclusion Criteria:

1. Greater than (>) 18 years
2. Considered by the treating physician for lenvatinib/pembolizumab combination therapy for the approved indications in Korea, prior to study
3. Provided written consent for use of personal medical information for the study purpose
4. Meets the approved indication and none of the contraindications for lenvatinib/pembrolizumab combination therapy in Korea, as confirmed by the treating physician

Exclusion Criteria:

1. Currently receiving lenvatinib and pembrolizumab as part of a clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean participants who are prescribed with lenvatinib in combination with pembrolizumab per the approved prescribing information will be enrolled in the study.
Sampling Method: Non-Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Serious Adverse Events (SAEs) | From the first dose of the study drug up to 48 weeks
  A SAE is defined as any untoward medical occurrence: resulting in death; life threatening requiring hospitalization or prolongation of hospitalization; resulting in persistent or significant disability or incapacity; resulting in birth defect or congenital anomaly or medically important due to other reasons than above mentioned criteria.
Number of Participants With Serious Adverse Drug Reactions (ADRs) | From the first dose of the study drug up to 48 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. Adverse events (AEs) with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Unexpected AEs | From the first dose of the study drug up to 48 weeks
  An AE is defined as any untoward and unintended signs (.example, anomalies in laboratory test results) or symptoms/diseases occurring during administration/use of drugs, etc., which do not necessarily have a causal relationship with the drug in question.
Number of Participants With Unexpected ADRs | From the first dose of the study drug up to 48 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Known ADRs | From the first dose of the study drug up to 48 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.
Number of Participants With Non-serious ADRs | From the first dose of the study drug up to 48 weeks
  An ADR is defined as harmful and unintended responses to the normal administration/use of drugs, in which a causal relationship with the drug in question cannot be ruled out. AEs with unknown causality to the drug among those voluntarily reported will be also considered ADRs.

SECONDARY OUTCOMES:
Percentage of Participants With a Best Overall Response (BOR) of Complete Response (CR), Partial Response (PR) and Stable Disease (SD) [Objective Response Rate (ORR)] | From the first dose of the study drug up to 48 weeks
  ORR is defined as the percentage of participants with BOR of CR, PR and SD as determined by investigator.

CONTACTS AND LOCATIONS:
Locations (19):
- South Korea (19):
  - Eisai Site #04, Bundang
  - Eisai Site #02, Busan
  - Eisai Site #10, Busan
  - Eisai Site #17, Busan
  - Eisai Site #06, Daegu
  - Eisai Site #03, Ilsan
  - Eisai Site #05, Jeonju
  - Eisai Site #08, Seoul
  - Eisai Site #09, Seoul
  - Eisai Site #11, Seoul
  - Eisai Site #12, Seoul
  - Eisai Site #13, Seoul
  - Eisai Site #14, Seoul
  - Eisai Site #15, Seoul
  - Eisai Site #16, Seoul
  - Eisai Site #19, Seoul
  - Eisai Site #21, Seoul
  - Eisai Site #22, Seoul
  - Eisai Site #23, Seoul

IPD SHARING:
Plan to Share IPD: Yes
Eisai's data sharing commitment and further information on how to request data can be found on our website http://eisaiclinicaltrials.com/.